CLINICAL TRIAL: NCT01279057
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group, Multi-Site Study to Compare the Clinical Equivalence of Fluticasone Furoate Nasal Spray (Lek Pharmaceuticals) With Veramyst® Nasal Spray (GlaxoSmithKline) in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Brief Title: A Study Comparing Two Fluticasone Furoate Nasal Sprays in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71047201
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Rhinitis; Seasonal Allergic Rhinitis; Fluticasone furoate; Equivalence; Hay fever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Fluticasone furoate 27.5 mcg/actuation nasal spray (Lek Pharmaceuticals) administered once daily at a dose of 110 mcg (4 actuations) for 14 days.
  Interventions: Drug: Fluticasone furoate 27.5 mcg/actuation nasal spray (Lek Pharmaceuticals)
- Reference (Active Comparator): Fluticasone furoate (Veramyst®) 27.5 mcg/actuation nasal spray administered once daily at a dose of 110 mcg (4 actuations) for 14 days.
  Interventions: Drug: Fluticasone furoate (Veramyst®) 27.5 mcg/actuation nasal spray
- Placebo (Placebo Comparator): Placebo nasal spray administered once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone furoate 27.5 mcg/actuation nasal spray (Lek Pharmaceuticals) — Nasal spray administered once daily at a dose of 110 mcg (4 actuations) for 14 days.
  Arms: Test
Drug: Fluticasone furoate (Veramyst®) 27.5 mcg/actuation nasal spray — Nasal spray administered once daily at a dose of 110 mcg (4 actuations) for 14 days.
  Arms: Reference
Drug: Placebo — Placebo nasal spray administered once daily (4 actuations) for 14 days.
  Arms: Placebo

SUMMARY:
This study compared the safety and efficacy of a generic fluticasone furoate (Lek Pharmaceuticals) nasal spray to the reference listed drug in the treatment of seasonal allergic rhinitis. Additionally both the test and the reference formulations were tested for superiority against a placebo nasal spray.

DETAILED DESCRIPTION:
The study was designed as a double-blind, randomized, placebo-controlled, parallel group, multi-site to compare the clinical equivalence of the test formulation of fluticasone furoate, 27.5 mcg/actuation nasal spray (Lek Pharmaceuticals d.d.) with the reference formulation Veramyst® nasal spray (GlaxoSmithKline) in the relief of the signs and symptoms of seasonal allergic rhinitis. Participants who met the inclusion/exclusion criteria entered a 7-day placebo lead-in period. Following this placebo lead-in period, on Day 1 participants who continued to meet eligibility criteria were randomly assigned in a 2:2:1 ratio to one of three treatment groups (Test Product:Reference Product:Placebo) for 14 days of treatment. In all treatment groups, participants were instructed to administer the study drug once daily at approximately the same time each day. A single dose of 110 mcg was 4 actuations, each containing 27.5 mcg per actuation. Patients were instructed to administer the 4 actuations alternating between right and left nostril, such that 2 actuations were not administered back to back to the same nostril.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 12 years of age or older with a minimum of 2 years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* Signed informed consent (assent) form.
* Documented positive allergic skin test to local pollen.
* An average score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) with a minimum score of at least 2 for "nasal congestion" and at least 4 on the reflective Total Ocular Symptom Score (rTOSS).

Exclusion Criteria:

* History of asthma that required chronic therapy (with the exception of occasional acute or mild exercise induced asthma).
* Some other past and concomitant medical conditions, prohibited medications.
* Upper respiratory tract infection or any untreated infections.
* Patient has started immunotherapy/changed the dose.
* Any known allergy to any of the components of the study nasal spray.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 727 (Actual)
Dates: Start 2010-12-27 (Actual); Primary Completion 2011-02-08 (Actual); Study Completion 2011-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Sandoz Investigational Site, Austin, Texas
  - Sandoz Investigational Site, Kerrville, Texas
  - Sandoz Investigational Site, New Braunfels, Texas
  - Sandoz Investigational Site, San Antonio, Texas
  - Sandoz Investigational Site, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 10 investigative sites in 1 country.
Pre-assignment Details: Participants who met the inclusion/exclusion criteria entered a 7-day placebo lead-in period. Following this placebo lead-in period, on Day 1 participants who continued to meet eligibility criteria were randomly assigned in a 2:2:1 ratio to one of three treatment groups (Test Product:Reference Product:Placebo).
Period: Overall Study
Arm/Group | Test | Reference | Placebo
Started | 288 | 292 | 147
Per-Protocol (PPP) Population (All participants who satisfied the criteria set forth in the protocol in terms of dosing compliance, number of available post-randomization evaluations and absence of significant protocol violations.) | 257 | 245 | 126
Intent-to-Treat (ITT) Population (All participants in the PPP as well as all participants who administered at least one dose of randomized study drug and had at least one post-randomization evaluation.) | 284 | 285 | 144
Completed | 282 | 287 | 144
Not Completed | 6 | 5 | 3
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Insufficient therapeutic response | 0 | 0 | 1
Not completed — Restricted medication for seasonal allergic rhinitis | 0 | 1 | 0
Not completed — Withdrew consent | 2 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Other | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 288 | 292 | 147 | 727
Age, Customized [Count of Participants; unit: Participants]
  < 18 | 17 | 28 | 17 | 62
  18 - 40 | 133 | 122 | 65 | 320
  41 - 64 | 122 | 137 | 59 | 318
  65 - 75 | 15 | 4 | 6 | 25
  > 75 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 195 | 91 | 460
  Male | 114 | 97 | 56 | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 233 | 241 | 126 | 600
  Black/African American | 50 | 40 | 19 | 109
  Asian | 2 | 5 | 2 | 9
  Native Hawaiian / Other Pacific Islander | 0 | 2 | 0 | 2
  American Indian / Alaska Native | 2 | 0 | 0 | 2
  Other | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: PRIMARY: Mean Change From Baseline in Reflective Total Nasal Symptom Score (rTNSS) (Equivalence: Per-Protocol Population)
Description: Patients were required to record a 12 hour "reflective" score twice a day approximately 12 hours apart. For the rTNSS patients were asked to "look back" or "reflect" on their severity of nasal symptoms over the previous 12 hours. The first rating on each day was taken prior to dosing. Patients were asked to score 4 nasal symptoms (nasal congestion, runny nose, sneezing and itchy nose) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 4 individual symptom scores obtained over the randomized treatment period were summed to give the mean rTNSS, which ranged from 0 to 12 with a lower score indicating less severe symptoms.
  Mean baseline rTNSS was calculated by summing the means of the 4 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline rTNSS" - "mean post-randomization rTNSS". A positive change from baseline in rTNSS is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: Per-Protocol population was used in this analysis. To determine equivalence, only the test and reference treatment arms were analyzed.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 257 | 245
score on scale | 2.036 (2.415) | 1.904 (2.409)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — If the 90% confidence intervals were contained within the interval 80.0% to 125.0%, then the two products were considered to be therapeutically equivalent; Ratio Test/Ref. Least Squares (LS) Means = 104.085, 90% CI 2-sided [87.421 to 124.210]

2. Primary Outcome: PRIMARY: Mean Change From Baseline in Reflective Total Nasal Symptom Score (rTNSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 1
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 284 | 284 | 144
score on scale | 2.035 (2.362) | 1.845 (2.378) | 0.952 (1.842)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA

3. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (iTNSS) (Equivalence: Per-Protocol Population)
Description: Participants were required to record an "instantaneous" score twice a day approximately 12 hours apart. For the iTNSS participants were asked to evaluate "how I feel now" regarding their severity of nasal symptoms. The first rating on each day was taken prior to dosing. Participants were asked to score 4 nasal symptoms (nasal congestion, runny nose, sneezing and itchy nose) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 4 individual symptom scores obtained over the randomized treatment period were summed to give the mean iTNSS, which ranged from 0 to 12 with a lower score indicating less severe symptoms.
  Mean baseline iTNSS was calculated by summing the means of the 4 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline iTNSS" - "mean post-randomization iTNSS". A positive change from baseline in iTNSS is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 257 | 245
score on scale | 2.017 (2.439) | 1.854 (2.411)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% confidence intervals within the interval 80.0% to 125.0%; Ratio Test/Ref. LS Means = 106.635, 90% CI 2-sided [89.256 to 127.790]

4. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (iTNSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 3
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 284 | 284 | 144
score on scale | 1.994 (2.398) | 1.805 (2.398) | 0.846 (1.981)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

5. Secondary Outcome: Mean Change From Baseline in Reflective Total Ocular Symptom Score (rTOSS) (Equivalence: Per-Protocol Population)
Description: Patients were required to record a 12 hour "reflective" score twice a day approximately 12 hours apart. For the rTOSS patients were asked to "look back" or "reflect" on their severity of ocular symptoms over the previous 12 hours. The first rating on each day was taken prior to dosing. Patients were asked to score 3 ocular symptoms (eye redness, itching/burning eyes, and tearing/watering eyes) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 3 individual symptom scores obtained over the randomized treatment period were summed to give the mean rTOSS, which ranged from 0 to 9 with a lower score indicating less severe symptoms.
  Mean baseline rTOSS was calculated by summing the means of the 3 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline rTOSS" - "mean post-randomization rTOSS". A positive change from baseline is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 257 | 245
score on scale | 1.388 (1.831) | 1.152 (1.790)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% confidence intervals within the interval 80.0% to 125.0%; Ratio Test/Ref. LS Means = 115.877, 90% CI 2-sided [94.129 to 143.949]

6. Secondary Outcome: Mean Change From Baseline in Reflective Total Ocular Symptom Score (rTOSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 5
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 284 | 284 | 144
score on scale | 1.373 (1.795) | 1.128 (1.762) | 0.787 (1.527)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0018, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0441, ANCOVA

7. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Ocular Symptom Score (iTOSS) (Equivalence: Per-Protocol Population)
Description: Patients were required to record an "instantaneous" score twice a day approximately 12 hours apart. For the iTOSS patients were asked to evaluate "how I feel now" regarding their severity of ocular symptoms. The first rating on each day was taken prior to dosing. Patients were asked to score 3 ocular symptoms (eye redness, itching/burning eyes, and tearing/watering eyes) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 3 individual symptom scores obtained over the randomized treatment period were summed to give the mean rTOSS, which ranged from 0 to 9 with a lower score indicating less severe symptoms.
  Mean baseline rTOSS was calculated by summing the means of the 3 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline iTOSS" - "mean post-randomization iTOSS". A positive change from baseline in iTOSS is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 257 | 245
score on scale | 1.389 (1.884) | 1.135 (1.803)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% confidence intervals within the interval 80.0% to 125.0%; Ratio Test/Ref. LS Means = 117.712, 90% CI 2-sided [95.410 to 146.583]

8. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Ocular Symptom Score (iTOSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 7
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 284 | 284 | 144
score on scale | 1.362 (1.851) | 1.118 (1.784) | 0.787 (1.563)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0018, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0451, ANCOVA

ADVERSE EVENTS:
Time Frame: From first dose of randomized treatment until last dose plus 1-4 days (up to Day 15 + 3).
Description: Any signs or symptoms that occurs during randomized treatment period plus the 1-4 days post treatment.
Arm/Group | Test | Reference | Placebo
All-Cause Mortality (participants affected / at risk) | 0/288 | 0/292 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/288 | 0/292 | 1/147
Other Adverse Events (participants affected / at risk) | 6/288 | 4/292 | 4/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=288) | Reference (N=292) | Placebo (N=147)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=288) | Reference (N=292) | Placebo (N=147)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.